CLINICAL TRIAL: NCT05908188
Title: Analysis of Mandibular Movements to Optimize Ventilatory Management of Children With Obstructive Sleep Apnea Syndrome Treated With Continuous Positive Airway Pressure or Non-Invasive Ventilation.
Brief Title: Analysis of Mandibular Movements in Ventilated Children With Sleep Apnea Syndrome
Acronym: AMANDA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A02697-34
Record Dates: First submitted 2021-12-20; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-02

CONDITIONS: Apnea Syndrome; Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; apnea syndrome; children; continuous positive pressure; non invasive ventilation
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obstructive Sleep Apnea is a common medical condition in children. Diagnosis is based on polysomnography . We conducted an open prospective non randomised clinical trial to assess the efficacy of a new medical device called SUNRISE.

DETAILED DESCRIPTION:
Obstructive Sleep apnea affects 4 percent of children. The standard device for the diagnosis and follow up is the polysomnography (PSG). However acess for this technique is difficult and expensive in certain institutions . Moreover, not all centers are qualified to receive the pediatric population. Thus expert consensus is present on the need for the development of a less expensive and easily accessible device to ensure the equality in medical care.

Recently an innovative medical device utilising the artificial intelligence technology is used to diagnose OSA in adults by recording the mandibular movement. Martinot et al were the first to use this device in children and noted a correlation between the mandibular movements and polysomnography measurements.

A multidisciplinary approach is used in the treatment of OSA. Indeed, the treatment is based on continous positive pressure and non invasive ventilation. To better evaluate the treatment, the sensor can be an alternative allowing to analyze the mandibular movements without moving at home.

We conducted an open prospective non randomised clinical trial to assess the efficacy of a new medical device called "SUNRISE" in the diagnosis and monitoring of OSA.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-18 years inclusive.
* With a diagnosis of severe OSA diagnosed at PSG, defined by an apnoea-hypopnoea index ≥ 10/ hours or an apnoea index ≥ 5/ hours, and associated or not with alveolar hypoventilation.
* Ventilated with noninvaisve ventilation or continuous positive airway pressure during sleep.
* With a nasal or nostril interface.
* Followed in one of the 2 participating centres: the Grenoble-Alpes University Hospital or the Trousseau Hospital in Paris.

Exclusion Criteria:

* Patients with centrally-induced sleep apnoea syndrome.
* Patients at the end of life or for whom limitation of active therapies has been established.
* Patients ventilated with a naso-oral interface.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: My population consists of children aged between 5 and 18 years old with obstructive sleep apnea syndrome and treated with positive pressure ventilation and non invasive ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Concomitant detection of residual obstructive breathing events by mandibular movements recorded by the sensor in comparison with a complete polysomnography recording performed in hospital under continuous positive pressure or non invasive ventilation | 1 year
  during one night in hospital and one night at home

SECONDARY OUTCOMES:
Residual obstructive airway events detected by mandibular movements and integrated continuous positive pressure or non invasive ventilation monitoring software. | 1 year
  the number of apnea and obstructive hypopnea per hour
The Obstructive Respiratory disturbance Index (ORDI) reproductibility | 1 year
  To compare the Obstructive Respiratory disturbance Index (ORDI) (defined as the number of obstructive apneas, hypopneas, and flow limitation events per hour) calculated during the hospital recording and that calculated during the home recording.
The difference in the Obstructive Respiratory disturbance Index (ORDI) before and after the modification of ventilatory parameters | 1 year
  The difference between the ORDI ((defined as the number of obstructive apneas, hypopneas, and flow limitation events per hour) at hospital recording and at home recording.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Mortamet, MD, Principal Investigator — Grenoble Alpes University Hospital
Locations (1):
- Grenoble University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaditis AG, Alonso Alvarez ML, Boudewyns A, Alexopoulos EI, Ersu R, Joosten K, Larramona H, Miano S, Narang I, Trang H, Tsaoussoglou M, Vandenbussche N, Villa MP, Van Waardenburg D, Weber S, Verhulst S. Obstructive sleep disordered breathing in 2- to 18-year-old children: diagnosis and management. Eur Respir J. 2016 Jan;47(1):69-94. doi: 10.1183/13993003.00385-2015. Epub 2015 Nov 5. PMID 26541535
- [Background] Lescanne E, Chiron B, Constant I, Couloigner V, Fauroux B, Hassani Y, Jouffroy L, Lesage V, Mondain M, Nowak C, Orliaguet G, Viot A; French Society of ENT (SFORL); French Association for Ambulatory Surgery (AFCA); French Society for Anaesthesia, Intensive Care (SFAR). Pediatric tonsillectomy: clinical practice guidelines. Eur Ann Otorhinolaryngol Head Neck Dis. 2012 Oct;129(5):264-71. doi: 10.1016/j.anorl.2012.03.003. Epub 2012 Oct 15. PMID 23078979
- [Background] Redline S, Tishler PV, Schluchter M, Aylor J, Clark K, Graham G. Risk factors for sleep-disordered breathing in children. Associations with obesity, race, and respiratory problems. Am J Respir Crit Care Med. 1999 May;159(5 Pt 1):1527-32. doi: 10.1164/ajrccm.159.5.9809079. PMID 10228121
- [Background] Aubertin G, Schroder C, Sevin F, Clouteau F, Lamblin MD, Vecchierini MF. [Obstructive sleep apnea-hypopnea syndrome in children: Clinical diagnosis]. Arch Pediatr. 2017 Feb;24 Suppl 1:S7-S15. doi: 10.1016/j.arcped.2016.09.002. Epub 2016 Oct 18. French. PMID 27769627
- [Background] Abrahamyan L, Sahakyan Y, Chung S, Pechlivanoglou P, Bielecki J, Carcone SM, Rac VE, Fitzpatrick M, Krahn M. Diagnostic accuracy of level IV portable sleep monitors versus polysomnography for obstructive sleep apnea: a systematic review and meta-analysis. Sleep Breath. 2018 Sep;22(3):593-611. doi: 10.1007/s11325-017-1615-1. Epub 2018 Jan 9. PMID 29318566
- [Background] Uddin MB, Chow CM, Su SW. Classification methods to detect sleep apnea in adults based on respiratory and oximetry signals: a systematic review. Physiol Meas. 2018 Mar 26;39(3):03TR01. doi: 10.1088/1361-6579/aaafb8. PMID 29446755
- [Background] Lapina VA, Dontsov AE, Ostrovskii MA, Emanuel' NM. [Interaction of oxygen anion radicals with eye melanins and ommochromes]. Dokl Akad Nauk SSSR. 1985;280(6):1463-5. No abstract available. Russian. PMID 2985349
- [Background] Gray EL, Barnes DJ. Beyond the thermistor: Novel technology for the ambulatory diagnosis of obstructive sleep apnoea. Respirology. 2017 Apr;22(3):418-419. doi: 10.1111/resp.13004. Epub 2017 Feb 14. No abstract available. PMID 28198129
- [Background] Obermeyer Z, Emanuel EJ. Predicting the Future - Big Data, Machine Learning, and Clinical Medicine. N Engl J Med. 2016 Sep 29;375(13):1216-9. doi: 10.1056/NEJMp1606181. No abstract available. PMID 27682033
- [Background] Amaddeo A, Caldarelli V, Fernandez-Bolanos M, Moreau J, Ramirez A, Khirani S, Fauroux B. Polygraphic respiratory events during sleep in children treated with home continuous positive airway pressure: description and clinical consequences. Sleep Med. 2015 Jan;16(1):107-12. doi: 10.1016/j.sleep.2014.07.030. Epub 2014 Nov 18. PMID 25541022
- [Background] Pepin JL, Letesson C, Le-Dong NN, Dedave A, Denison S, Cuthbert V, Martinot JB, Gozal D. Assessment of Mandibular Movement Monitoring With Machine Learning Analysis for the Diagnosis of Obstructive Sleep Apnea. JAMA Netw Open. 2020 Jan 3;3(1):e1919657. doi: 10.1001/jamanetworkopen.2019.19657. PMID 31968116
- [Background] Martinot JB, Senny F, Denison S, Cuthbert V, Gueulette E, Guenard H, Pepin JL. Mandibular movements identify respiratory effort in pediatric obstructive sleep apnea. J Clin Sleep Med. 2015 Apr 15;11(5):567-74. doi: 10.5664/jcsm.4706. PMID 25766710
- [Background] Berry RB, Budhiraja R, Gottlieb DJ, Gozal D, Iber C, Kapur VK, Marcus CL, Mehra R, Parthasarathy S, Quan SF, Redline S, Strohl KP, Davidson Ward SL, Tangredi MM; American Academy of Sleep Medicine. Rules for scoring respiratory events in sleep: update of the 2007 AASM Manual for the Scoring of Sleep and Associated Events. Deliberations of the Sleep Apnea Definitions Task Force of the American Academy of Sleep Medicine. J Clin Sleep Med. 2012 Oct 15;8(5):597-619. doi: 10.5664/jcsm.2172. PMID 23066376
- [Background] Amaddeo A, Frapin A, Touil S, Khirani S, Griffon L, Fauroux B. Outpatient initiation of long-term continuous positive airway pressure in children. Pediatr Pulmonol. 2018 Oct;53(10):1422-1428. doi: 10.1002/ppul.24138. Epub 2018 Aug 1. PMID 30070059
- [Background] Amaddeo A, Frapin A, Fauroux B. Long-term non-invasive ventilation in children. Lancet Respir Med. 2016 Dec;4(12):999-1008. doi: 10.1016/S2213-2600(16)30151-5. Epub 2016 Jul 13. PMID 27423917
- [Background] Amaddeo A, Khirani S, Griffon L, Teng T, Lanzeray A, Fauroux B. Non-invasive Ventilation and CPAP Failure in Children and Indications for Invasive Ventilation. Front Pediatr. 2020 Oct 26;8:544921. doi: 10.3389/fped.2020.544921. eCollection 2020. PMID 33194886